CLINICAL TRIAL: NCT06683274
Title: Bascom Cleft Lift for Primary Wound Healing in Complex and Recurrent Sacrococcygeal Pilonidal Sinus Disease
Acronym: BATCRAC
Status: Recruiting | Type: Observational
Sponsor: Albert Schweitzer Ziekenhuis, Netherlands (Other)
Responsible Party: Principal Investigator, Max Goudberg, MD, PhD candidate, Albert Schweitzer Ziekenhuis, Netherlands
Other Study IDs: 2024.077; 2024.077 (Other: ASz)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pilonidal Sinus
Keywords: Pilonidal sinus; Bascom cleft lift
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control cohort: Current practice cohort
- Interventional cohort: Best practice care pathway with standardized Bascom cleft lift

SUMMARY:
The goal of this observational study is to improve care for patients with complex or recurrent pilonidal sinus disease by developing and implementing a best practice care pathway, including a standardized cleft lift operation.

The main question it aims to answer is: Does a best practice care pathway with standardized cleft lift operation lead to shorter wound healing time and time to return to normal activities, compared to current standard care, with traditional excision techniques.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age and older
* Symptomatic complex or recurrent pilonidal sinus disease
* Planned for surgical treatment
* Signed informed consent

Exclusion Criteria:

* Pregnant
* Insufficient understanding of the Dutch language or otherwise unable to give consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with (symptomatic) complex or recurrent pilonidal sinus disease, who will be planned for surgical treatment.
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | The outcome will be evaluated at each follow-up visit, at 1-3 weeks, 4-6 weeks and 6 months postoperative. If necessary, additional visits will be planned
  Time to wound healing (in days), this will be self reported by patients when the skin is completely closed, and will be validated through clinical assessment by the surgeon.

SECONDARY OUTCOMES:
Return to normal activities | The outcome will be evaluated at each follow-up visit, at 1-3 weeks, 4-6 weeks and 6 months postoperative. If necessary, additional visits will be planned
  Time to return to normal activities after surgery (in days). This will be self reported by patients through a brief checklist on which the activities (washing, dressing, sitting, work/study) should be checked when possible without discomfort.

OTHER OUTCOMES:
Quality of Life | Baseline, 4-6 weeks and 6 months postoperative.
  Quality of Life, measured with EuroQol 5 dimensions, 5 levels (EQ-5D-5L) questionnaire. The questions are answered on a 5 point Likert scale. Ranging from 5-25, with 5 being the best possible outcome and 25 being the worst possible outcome. Additionally, there is a general question on a 0-100 scale, with 0 being the worst health possible and 100 being the best health possible.
Pain | The outcome will be evaluated at each follow-up visit, at 1-3 weeks, 4-6 weeks and 6 months postoperative.
  Pain score, on a Numeric Rating Scale ranging from 0-10 with 0 representing 'no pain' and 10 representing 'the worst pain possible'

CONTACTS AND LOCATIONS:
Overall Officials: Robert Smeenk, MD, PhD, Principal Investigator — Albert Schweitzer Ziekenhuis, Netherlands; Boudewijn Toorenvliet, MD, PhD, Principal Investigator — Ikazia ziekenhuis
Locations (1):
- Albert Schweitzer ziekenhuis, Dordrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No